CLINICAL TRIAL: NCT01796730
Title: A 12-week, Double-blind, Multicenter, 3-crossover, Placebo Controlled and Randomized Trial to Investigate the Efficacy and Safety of 10mg and 5mg Bambuterol Tablets Once Daily in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effects and Safety of Different Dose of Bambuterol on Chinese COPD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, jingping Zheng, Vice Director of Guangzhou Institution of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIRDBAM201201
Record Dates: First submitted 2013-02-05; First posted 2013-02-22 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: COPD
Keywords: efficacy; safety; Bambuterol tablets; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — bambuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sequence I (Experimental): 10mg (21 days) -washout (7 days) - bambuterol 5mg (21 days) -washout (7 days) -placebo (21 days)
  Interventions: Drug: bambuterol; Drug: Placebo
- sequence II (Experimental): bambuterol 5mg (21 days) -washout (7 days) - placebo (21 days) -washout (7 days) - bambuterol 10mg (21 days)
  Interventions: Drug: bambuterol; Drug: Placebo
- sequence III (Experimental): placebo (21 days) -washout (7 days) - bambuterol 10mg (21 days) - washout (7 days) - bambuterol 5mg (21 days)
  Interventions: Drug: bambuterol; Drug: Placebo

INTERVENTIONS:
Drug: bambuterol — Patients will be randomized allocated to receive three treatment sequences I, II and III, every treatment period is separated by a washout period of 7 days.
  Other Names: Bambec, KWD-2183
Drug: Placebo

SUMMARY:
This is a randomized, double-blind, 3-crossover trial with a 7-days washout baseline period followed by three treatment periods of 21-days each performed in patients with COPD. Patients will be randomized to receive three treatments (bambuterol 10mg, bambuterol 5 mg and placebo).

DETAILED DESCRIPTION:
Patients with COPD who meet the inclusion criteria will enter the 7-days washout baseline period. After the baseline period, patients will be randomly assigned to one of the following treatment sequences:

* Sequence I: bambuterol 10mg (21 days) -washout (7 days) - bambuterol 5mg (21 days) - washout (7 days) - placebo (21 days);
* Sequence II: bambuterol 5mg (21 days) -washout (7 days) - placebo (21 days) - washout (7 days) - bambuterol 10mg (21 days) ;
* Sequence III: placebo (21 days) -washout (7 days) - bambuterol 10mg (21 days) - washout (7 days) - bambuterol 5mg (21 days).

During the treatment period patients will record their adverse events and use of rescue medication (Ipratropium bromide) in a diary. At each visit, pulmonary function tests will be performed. At V2, V4 and V6, forced expiratory volume at one second (FEV1) and forced vital capacity (FVC) are measured at following times: immediately before tablet treatment, and at 0.5, 1, 2, 3, 4, 6, 9, 12hrs after administration of tablets, FEV1 and FVC area under curve (AUC) 0~12 hours will be analyzed. At V1, V3, V5 and V7, and FVC are measured a time in the morning. Peak expiratory flow rate (PEFR) is measured by Mini-Wright peak flow meter in the morning before treatments. All other data will be evaluated as safety status, and monitoring of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* COPD, the disease is under a stable phase
* Giving written informed consent
* Age 40 - 80 years (both inclusive)
* Chinese ethnicity
* 30% of predicated normal ≤Post bronchodilator FEV1 ≤ 70% of predicated normal
* Post bronchodilator FEV1/FVC ≤ 70% (Note: post bronchodilator FEV1 will be tested 20-30 minutes after Salbutamol is used (inhaled via metered dose inhaler (MDI) and spacer).

Exclusion Criteria:

* COPD acute exacerbation 4 weeks prior to the enrollment
* Patients with a history of asthma, allergic rhinitis, atopy
* Use of disallowed drugs
* Clinically relevant abnormal laboratory values suggesting an undiagnosed disease requiring further clinical evaluation (as assessed by the Investigator)
* Severe psychiatric or neurological disorders
* Congestive heart failure severity grade IV according to New York Heart Association (NYHA)
* Haemodynamically significant cardiac arrhythmias or heart valve deformations
* CT or X-ray findings indicating an acute pulmonary disease other than COPD (e.g. tuberculosis, severe bronchiectasis, tumors)
* Severe immunological diseases (e.g. HIV infection, multiple sclerosis, lupus erythematosus, progressive multifocal leukoencephalopathy)
* Severe acute infectious diseases (e.g. tuberculosis or acute hepatitis)
* Any diagnosis of a malignant disease (except basal cell carcinoma) within 5 years before trial start
* Alcohol or drug abuse within the past year
* Suspected hypersensitivity to the Bambuterol or ingredients thereof, or any other contraindication for the use thereof
* Pregnancy, breast feeding, planned oocyte donation or oocyte implantation
* Participation in another trial (use of investigational product) within 30 days preceding the baseline visit V1 or re-entry of patients previously enrolled in this trial
* Suffering from any concomitant disease that might interfere with trial procedures or evaluations

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
the change in FEV1(L) and FVC(L) | pre- and post-treatment during 0 to 3 week, 4 to 7 week and 8 to 11 week
  The primary endpoints will be the difference in FEV1 as well as FVC between pre-treatment and post-treatment at respective treatment period (ie. Visit 2(0 week) and Visit 3(3 week), Visit 4 (4 week)and Visit 5(7 week), Visit 6 (8 week) and Visit 7(11 week)) .

SECONDARY OUTCOMES:
difference of AUC(0-12h) FEV1(L) as well as AUC(0-12h) FVC(L) among 3 dose groups | at 0, 4, 8 week
  * AUC FEV1: 0-12h in V2 (0 week), V4 (4 week) and V6 (8 week),
  * AUC FVC: 0-12h in V2 (0 week), V4 (4 week) and V6 (8 week),
change of PEFR(L/min) | during 0 to 3 week, 4 to 7 week and 8 to 11 week
  difference of Peak flow rate (PEFR) during the treatment period among 3 dose groups

OTHER OUTCOMES:
use of rescue medication | during 0 to 3week,4 to 7 week and 8 to 11 week
  •difference of use of rescue medication (Ipratropium bromide) during the treatment period among 3 dose groups
The Baseline Dyspnea Index (BDI) and Transition Dyspnoea Index (TDI) | BDI at 0, 4 and 8 week, TDI at 3, 7 and 11 week
  The Baseline Dyspnea Index (BDI) will be collected before each treatment period, ie. at visits of 2, 4, 6.
  Transition Dyspnoea Index (TDI) will be collected at the end of each treatment period, ie. at visits of 3, 5, 7.
Tremor, Palpitation | up to 11 weeks
  Difference of frequency and severity of tremor, palpitation and other adverse events among 3 dose groups will be collected and analyzed during the whole study period.
electrocardiogram (ECG) | at -1,0,3,4,7,8,11 week
  Electrocardiogram (ECG) will be assessed at all visits

CONTACTS AND LOCATIONS:
Overall Officials: Jinping Zheng, MD, Principal Investigator — Guagnzhou Institute of Respiratory Disease, First affiliated hospital of Guangzhou Medical University
Locations (3):
- China (3):
  - Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou Institution of Respiratory Disease (GIRD), The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong

REFERENCES:
- [Background] McDonald CF, Pierce RJ, Thompson PJ, Allen D, Bowler S, Breslin AB, Bowes G, Saunders N, Murree-Allen K, Frith P, Musk AW. Comparison of oral bambuterol and terbutaline in elderly patients with chronic reversible airflow obstruction. J Asthma. 1997;34(1):53-9. doi: 10.3109/02770909709071203. PMID 9033440
- [Background] Cazzola M, Calderaro F, Califano C, Di Pema F, Vinciguerra A, Donner CF, Matera MG. Oral bambuterol compared to inhaled salmeterol in patients with partially reversible chronic obstructive pulmonary disease. Eur J Clin Pharmacol. 1999 Jan;54(11):829-33. doi: 10.1007/s002280050561. PMID 10027655